CLINICAL TRIAL: NCT03126344
Title: Comparison King Vision Video Laryngoscopy 、McGrath MAC Video Laryngoscopy With Macintosh Laryngoscopy for Nasal Intubation
Brief Title: Nasal Intubation Using King Vision Video Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: suny2
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Nasal Intubation
Keywords: King Vision

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- King Vision video laryngoscope (Experimental)
  Interventions: Device: King Vision video laryngoscope
- McGrath MAC video laryngoscope (Experimental)
  Interventions: Device: McGrath MAC video laryngoscope
- Macintosh (Active Comparator)
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: King Vision video laryngoscope — nasal intubation using King Vision video laryngoscope Device after general anesthesia induction
  Arms: King Vision video laryngoscope
Device: McGrath MAC video laryngoscope — nasal intubation using McGrath MAC video laryngoscope Device after general anesthesia induction
  Arms: McGrath MAC video laryngoscope
Device: Macintosh laryngoscope — nasal intubation using Macintosh laryngoscope Device after general anesthesia induction
  Arms: Macintosh

SUMMARY:
This study was designed to determine the comparison between the King Vision video laryngoscope 、 McGrath MAC video laryngoscope and Macintosh laryngoscope for nasotracheal intubation.Patients were divided into 3 groups of 30 patients each.Patients of King Vision group [n=30]、 McGrath MAC group [n=30] and Macintosh group[n=30]were intubated using respective devices.This study is the first to search the use of King Vision video laryngoscope for nasotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* general anesthesia with nasotracheal intubation
* anticipated difficult airway

Exclusion Criteria:

* contraindications to nasal intubation
* Patients with a history of anti-hypertensive drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital,Affililated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu H, Liu J, Suo L, Zhou C, Sun Y, Jiang H. A randomized controlled comparison of non-channeled king vision, McGrath MAC video laryngoscope and Macintosh direct laryngoscope for nasotracheal intubation in patients with predicted difficult intubations. BMC Anesthesiol. 2019 Aug 31;19(1):166. doi: 10.1186/s12871-019-0838-z. PMID 31470814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh
Started | 33 | 33 | 33
Completed | 33 | 33 | 28
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 33 | 99
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 38 (12) | 36 (11) | 40 (11) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 16 | 50
  Male | 18 | 14 | 17 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 33 | 33 | 33 | 99
BMI [Mean (Standard Deviation); unit: Kg/M^2] | 22 (3) | 22 (3) | 22 (3) | 22 (3)
ASA I or II [Count of Participants; unit: Participants] — ASA I No organic,physiologic,biochemical or psychiatric disturbance ASA II A patient with mild systemic disease that reaults in no functional imitation.
  Participants | 33 | 33 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: the interval between opening the mouth and the time when three consecutive end-tidal CO2 waves were appeared on the monitor
Time Frame: 0 min after nasal intubation
Measure: Mean (Standard Deviation); unit: second
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh
Number analyzed (Participants) | 33 | 33 | 28
second | 37.6 (7.3) | 35.4 (8.8) | 46.8 (10.4)

2. Secondary Outcome: Laryngoscopy Time
Description: time to expose the glottis
Time Frame: after expose the glottis
Measure: Mean (Standard Deviation); unit: second
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh
Number analyzed (Participants) | 33 | 33 | 28
second | 16.7 (5.5) | 15.6 (6.3) | 22.8 (7.2)

3. Secondary Outcome: Number of Participants With Complications
Description: sore throat, hoarseness, etc
Time Frame: 24h after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh
Number analyzed (Participants) | 33 | 33 | 28
Participants | 6 | 7 | 21

ADVERSE EVENTS:
Time Frame: From the time of anesthesia induction to approximately 24 hours
Arm/Group | King Vision Video Laryngoscope | McGrath MAC Video Laryngoscope | Macintosh
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 6/33 | 9/33 | 21/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | King Vision Video Laryngoscope (N=33) | McGrath MAC Video Laryngoscope (N=33) | Macintosh (N=33)
bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
dental injury (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
soar throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 12 (12)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03126344/Prot_SAP_004.pdf
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03126344/ICF_005.pdf